CLINICAL TRIAL: NCT01533038
Title: BPH-6: A UroLift® System Post Market Multi-Center Randomized Study
Brief Title: BPH-6: Comparison of the UroLift System to TURP for Benign Prostatic Hyperplasia
Acronym: BPH-6
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NeoTract, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP12317
Record Dates: First submitted 2012-02-10; First posted 2012-02-15 (Estimated); Results first posted 2015-11-26 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-11

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- UroLift System (Active Comparator): UroLift System procedure
  Interventions: Device: UroLift System
- Transurethral Resection of the Prostate (Active Comparator): Transurethral Resection of the Prostate surgery
  Interventions: Procedure: Transurethral Resection of the Prostate

INTERVENTIONS:
Device: UroLift System — The NeoTract UroLift System is a medical device approved for sale in the European Union, Australia, New Zealand, Canada, Serbia, and Turkey. It was developed for the intended use of soft tissue approximation and for the treatment of lower urinary tract symptoms (LUTS) associated with Benign Prostatic Hyperplasia (BPH). During the procedure, an implant is delivered into the prostatic lobe obstructing the urethra and restricting urine flow. The distal end of the device is used to compress the lobe then the implant is delivered to retain the lobe in position, thereby increasing the urethral opening and reducing the fluid obstruction through the prostatic urethra.
  Arms: UroLift System
Procedure: Transurethral Resection of the Prostate — Transurethral Resection of the Prostate (TURP) is a surgical procedure which removes prostatic tissue by electrocautery dissection. During the procedure the tissue at the bladder neck and the adjacent adenoma are resected in quadrants. Resection continues into the midportion of the gland and concludes at the apex. Any remaining residual tissue is cleared, leaving a void from verumontanum to bladder neck.
  Arms: Transurethral Resection of the Prostate

SUMMARY:
The purpose of this study is to compare the UroLift System Treatment to Transurethral Resection of the Prostate (TURP) in improving a patient's overall quality of life, while evaluating healthcare expenditures associated with each therapy.

DETAILED DESCRIPTION:
The study is a prospective, consecutive, multi-center, 1:1 randomized study (UroLift System:TURP). The study is intended to be conducted at up to 20 different centers in Europe and Canada to enroll up to 100 subjects.

Subject follow-up visits are at 2 weeks, 1, 3, 6, 12 and 24 months for all subjects.

ELIGIBILITY:
Inclusion Criteria:

• Men >50 years old with moderate-severe BPH

Exclusion Criteria:

* Size, width of prostate
* Other medical condition or co-morbidity contraindicative for TURP or UroLift

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-02; Primary Completion 2015-10 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Montorsi, MD, Principal Investigator — University Vita Salute San Raffaele
Locations (9):
- Herlev Hospital, Herlev, Denmark
- Germany (4):
  - PAN Klinik, Cologne
  - University Hospital Freiburg, Freiburg im Breisgau
  - Ludwigs-Maximilians Universität / Klinikum Großhadern, Munich
  - University Hospital Tuebingen, Tübingen
- United Kingdom (4):
  - Frimley Park Hospital, Frimley
  - The Royal Hallamshire Hospital, Sheffield
  - City Hospitals Sunderland NHS Foundation Trust, Sunderland
  - Musgrove Park Hospital, Taunton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sonksen J, Barber NJ, Speakman MJ, Berges R, Wetterauer U, Greene D, Sievert KD, Chapple CR, Montorsi F, Patterson JM, Fahrenkrug L, Schoenthaler M, Gratzke C. Prospective, randomized, multinational study of prostatic urethral lift versus transurethral resection of the prostate: 12-month results from the BPH6 study. Eur Urol. 2015 Oct;68(4):643-52. doi: 10.1016/j.eururo.2015.04.024. Epub 2015 Apr 30. PMID 25937539

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | UroLift System | Transurethral Resection of the Prostate
Started | 45 | 35
Completed | 45 | 34
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | UroLift System | Transurethral Resection of the Prostate | Total
Number analyzed (Participants) | 45 | 35 | 80
Age, Customized [Mean (Full Range); unit: years]
  Age | 63 [49 to 84] | 65 [51 to 78] | 65 [49 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 45 | 35 | 80
Region of Enrollment [Number; unit: participants]
  Denmark | 10 | 9 | 19
  United Kingdom | 18 | 13 | 31
  Germany | 17 | 13 | 30

OUTCOME MEASURES:

1. Primary Outcome: Responder Analysis: A Subject is a Responder at the 12 Month Follow-up Time Point if All 6 Thresholds of the BPH-6 Endpoint Are Met
Description: 1. LUTS: ≥ 30% reduction in IPSS compared to baseline
  2. Recovery Experience: Return to pre-operative activity levels by 1 month
  3. Erectile function: Less than 6-point reduction in SHIM compared to baseline.
  4. Ejaculatory function: Response on MSHQ-EjD that indicates emission of semen. This excludes the response "Could not ejaculate"
  5. Continence: ISI score of 4 points or less at all follow-up time points
  6. Safety: No procedure-related adverse event greater than Grade I on the Clavien-Dindo classification system modified for TURP at any time during procedure or follow up.
Time Frame: Month 12
Measure: Number; unit: % Responders of Participants
Arm/Group | UroLift System | Transurethral Resection of the Prostate
Number analyzed (Participants) | 43 | 35
% Responders of Participants | 52 | 20

ADVERSE EVENTS:
Time Frame: SAEs Adjudication through 12M; AEs through 24M-(2 years post-Index)
Arm/Group | UroLift System | Transurethral Resection of the Prostate
Serious Adverse Events (participants affected / at risk) | 2/45 | 4/35
Other Adverse Events (participants affected / at risk) | 33/45 | 28/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UroLift System (N=45) | Transurethral Resection of the Prostate (N=35)
Weak urinary stream (Gastrointestinal disorders) | 1 (1) | 0 (0)
Blood clot in urine (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urge incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urethral Stricture (Gastrointestinal disorders) | 0 (0) | 1 (1)
Epididymitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Incomplete Bladder Empyting (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UroLift System (N=45) | Transurethral Resection of the Prostate (N=35)
Bladder spasm (Gastrointestinal disorders) | 1 (1) | 2 (2)
Bladder Tamponade (Gastrointestinal disorders) | 1 (1) | 1 (1)
Blood clot in urine (Gastrointestinal disorders) | 10 (10) | 15 (15)
Dysuria (Gastrointestinal disorders) | 17 (17) | 19 (19)
Epidymitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Erectile Dysfunction (Gastrointestinal disorders) | 0 (0) | 3 (3)
Hemaeturia (Gastrointestinal disorders) | 7 (7) | 6 (6)
Incomplete bladder empyting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Infection , urinary tract (Gastrointestinal disorders) | 4 (4) | 2 (3)
Lower urinary tract symptoms (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nocturia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pain, Abdominal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain, Groin (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pelvic Pain (Gastrointestinal disorders) | 5 (5) | 3 (3)
Post-void dribble (Gastrointestinal disorders) | 0 (0) | 2 (2)
Prostatic greenlight laser vaporization (Gastrointestinal disorders) | 0 (0) | 0 (0)
Prosthesis calcification (Gastrointestinal disorders) | 1 (1) | 0 (0)
Residual urine volume increase (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retrograde Ejaculation (Gastrointestinal disorders) | 0 (0) | 7 (7)
Stone, urinary bladder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Urge Incontinence (Gastrointestinal disorders) | 1 (1) | 6 (6)
Urinary Frequency (Gastrointestinal disorders) | 4 (4) | 4 (4)
Urinary urgency (Gastrointestinal disorders) | 5 (5) | 9 (9)
Weak urinary stream (Gastrointestinal disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No